CLINICAL TRIAL: NCT06092528
Title: Investigation of the Effects of Pulmonary Rehabilitation on Exercise Capacity, Muscle Oxygenation and Physical Activity Level in Children With Primary Immunodeficiency
Brief Title: Investigation of the Effects of Pulmonary Rehabilitation in Children With Primary Immunodeficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gazi University 73
Record Dates: First submitted 2023-09-28; First posted 2023-10-23 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Primary Immunodeficiency
Keywords: primary immunodeficiency; pulmonary rehabilitation; exercise capacity; muscle oxygenation; physical activity
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
  Evaluations and interventions will be performed different physiotherapist. In addition, before statistical analysis patients' groups will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): Pulmonary rehabilitation practices (inspiratory muscle training, aerobic exercise training, resistance exercise training) will be performed 3 sessions a week for 6 weeks under the supervision of a physiotherapist to the training group.
  Interventions: Other: Inspiratory muscle training; Other: Upper extremity aerobic exercise training; Other: Lower extremity aerobic exercise training; Other: Resistant exercise training
- Control Group (Sham Comparator): Control group will be given breathing exercises as a home program for 6 weeks.
  Interventions: Other: Thoracic expansion exercises

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training will be performed with Power Breathe®. Inspiratory muscle training will be given to the training group, starting from 50% of the MIP, and 2 sessions/day, 15 minutes/session. Patients will be asked to check breathing for 4-5 breaths after 8-10 consecutive breathing cycles. The patient will continue this cycle for 15 minutes.
  Arms: Pulmonary Rehabilitation Group
Other: Upper extremity aerobic exercise training — Upper extremity aerobic exercise training will be performed 3 days/week, 1 session/day, 15 min/session using arm ergometer device accompanied by a physiotherapist. Aerobic exercise training workload will be 60-80% of maximal heart rate. In this study, the perception of dyspnea will be between 3-4, arm fatigue and general fatigue perception will be between 5-6, warm-up and cool-down periods will be 5 minutes, and pedaling speed will be 40-50 rev/min, according to MBS.
  Arms: Pulmonary Rehabilitation Group
Other: Lower extremity aerobic exercise training — Lower extremity aerobic exercise training will be performed 3 days/week, 1 session/day, 15 minutes/session using the treadmill device, accompanied by a physiotherapist. Aerobic exercise training workload was set at 60-80% of maximal heart rate, dyspnea perception according to MBS was between 3-4, arm fatigue and general fatigue perception was between 5-6, and warm-up and cool-down periods were 5 minutes.
  Arms: Pulmonary Rehabilitation Group
Other: Resistant exercise training — Upper and lower additional limb strengthening training will be performed 3 days/week, 1 session/day, 10 repetitions/sessions from the first day by using bullion weights in the presence of a physiotherapist. The upper extremity strengthening program will consist of a progressive exercise program to strengthen the shoulder flexors and abductors, and the lower extremity strengthening program to strengthen the knee extensors. The training workload will be increased progressively. For strength training, the workload will be adjusted so that the perception of fatigue is between 4 and 6 according to MBS.
  Arms: Pulmonary Rehabilitation Group
Other: Thoracic expansion exercises — The control group will be asked to do thoracic expansion exercises seven days/week and 120 pieces/day for six weeks.
  Arms: Control Group

SUMMARY:
Primary immunodeficiencies (PID) are a heterogeneous group of diseases that occur as a result of disorders that affect the development, differentiation and/or function of various cells and building blocks in the immune system. Among the symptoms and complications of PID, pulmonary complications are very common and significantly increase the morbidity and mortality of the disease.

DETAILED DESCRIPTION:
Among the symptoms and complications of PID, pulmonary complications are very common and significantly increase the morbidity and mortality of the disease. Recurrent respiratory infections are often the first warning sign in some types of PID and is a cause of mortality in adults with PID. Presence of 2 or more pneumonias per year is one of the 10 warning signs of PID. Respiratory system diseases are mainly caused by acute and chronic infections. Non-infectious respiratory system diseases and complications are asthma, bronchiectasis, bronchiolitis obliterans, interstitial lung disease, granulomatous lung disease and malignancies. These diseases significantly affect the quality of life of PID patients, limiting their ability to work and their physical and social activities. Health-related quality of life in PID patients is also significantly affected by delays in the diagnosis and treatment of infections. As survival from infections increases, non-infectious pulmonary complications are more common in PID patients. Permanent lung damage is seen at a rate of 20-40%, especially in PID patients with antibody deficiency. The main causes of exercise intolerance in patients with lung disease include isolated or associated factors such as increased symptoms (fatigue and shortness of breath in the lower extremities), development of dynamic hyperinflation, peripheral muscle dysfunction, abnormalities in oxygen transport and progressive loss of physical condition, physical inactivity. There are no studies evaluating exercise capacity, respiratory and peripheral muscle strength, inspiratory muscle endurance, and muscle oxygenation in children with PID. In studies conducted with post-infectious bronchiolitis obliterans patients, it has been shown that exercise capacity is reduced in these patients. There are no studies in the literature on pulmonary rehabilitation practices and efficacy in PID patients.

The primary aim of this study: To investigate the effects of pulmonary rehabilitation on exercise capacity and muscle oxygenation in children with primary immunodeficiency.

The secondary aim of this study: To investigate the effects of pulmonary rehabilitation on physical activity level, respiratory functions, peripheral and respiratory muscle strength, inspiratory muscle endurance, shortness of breath, fatigue and quality of life in children with primary immunodeficiency.

Primary outcome measurement will be oxygen consumption (cardiopulmonary exercise test).

Secondary outcome will be muscle oxygenation (Moxy device), physical activity level (multi sensor activity device), pulmonary function (spirometer), functional exercise capacity (six-minute walk test), respiratory (mouth pressure device) and peripheral muscle (hand-held dynamometer) strength, inspiratory muscle endurance (incremental threshold loading test), dyspnea (Modified Borg Scale (MBS)), fatigue (Modified Borg Scale) and quality of life (The Pediatric Quality of Life Inventory (PedsQL)).

ELIGIBILITY:
Inclusion Criteria:

-Patients aged 6-18 years with primary immunodeficiency

Exclusion Criteria:

* Acute pulmonary exacerbation, acute upper or lower respiratory tract infection
* Serious neurological, neuromuscular, orthopedic and other systemic diseases or other diseases affecting physical functions
* Participating in a planned exercise program in the past three months
* Cognitive impairment, which may cause difficulty understanding and following exercise test instructions

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Oxygen Consumption | First Day
  Cardiopulmonary Exercises Test

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity (FVC)) | Second Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | Second Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | Second Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Second Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | Second Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, peak flow rate (PEF) will be evaluated.
Respiratory Muscle Strength | Second Day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria
Respiratory Muscle Endurance | Second Day
  Incremental threshold loading test
Peripheral Muscle Strength | Second Day
  Hand held dynamometer
Functional exercise capacity | Second Day
  6 minute walking test
Quality of Life (For Children) | First Day
  The Pediatric Quality of Life Inventory (PedsQL): It includes 8 items that measure physical functionality, 5 items that measure emotional functionality, 5 items that measure social functionality, and 5 items that assess functionality at school. There are separate forms for parents and children. There are separate scales for children 5-7 years old, 8-12 years old and 13-18 years old. For parents, there are separate forms for 2-4 years, 5-7 years, 8-12 years and 13-18 years. Items are scored between 0-100. The higher the total PedsQL score, the better the health-related quality of life is perceived.
Dyspnea | First and Second Day
  Modified Borg Scale: The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
Fatigue | First and Second Day
  Modified Borg Scale: The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
Muscle oxygenation | First and Second Day
  Moxy® monitor
Physical Activity Level (Total energy expenditure) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Active energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Physical activity time (min / day)will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Number of steps (steps / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Time spent lying down (min / day) days) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Sleep time (min / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yoleri, Pt. MsC, Principal Investigator — Gazi University; Caner Aytekin, Assoc. Prof., Principal Investigator — MH. Dr. Sami Ulus Children's Health and Diseases Training and Research Hospital; Meral Boşnak Güçlü, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Li AM, Yin J, Au JT, So HK, Tsang T, Wong E, Fok TF, Ng PC. Standard reference for the six-minute-walk test in healthy children aged 7 to 16 years. Am J Respir Crit Care Med. 2007 Jul 15;176(2):174-80. doi: 10.1164/rccm.200607-883OC. Epub 2007 Apr 26. PMID 17463419
- [Background] Crum EM, O'Connor WJ, Van Loo L, Valckx M, Stannard SR. Validity and reliability of the Moxy oxygen monitor during incremental cycling exercise. Eur J Sport Sci. 2017 Sep;17(8):1037-1043. doi: 10.1080/17461391.2017.1330899. Epub 2017 May 30. PMID 28557670
- [Background] Lee JA, Laurson KR. Validity of the SenseWear armband step count measure during controlled and free-living conditions. J Exerc Sci Fit. 2015 Jun;13(1):16-23. doi: 10.1016/j.jesf.2014.11.002. Epub 2015 Jan 29. PMID 29541094
- [Background] Patel SA, Benzo RP, Slivka WA, Sciurba FC. Activity monitoring and energy expenditure in COPD patients: a validation study. COPD. 2007 Jun;4(2):107-12. doi: 10.1080/15412550701246658. PMID 17530503
- [Background] Ridgers ND, Hnatiuk JA, Vincent GE, Timperio A, Barnett LM, Salmon J. How many days of monitoring are needed to reliably assess SenseWear Armband outcomes in primary school-aged children? J Sci Med Sport. 2016 Dec;19(12):999-1003. doi: 10.1016/j.jsams.2016.02.009. Epub 2016 Mar 3. PMID 26971298
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Domenech-Clar R, Lopez-Andreu JA, Compte-Torrero L, De Diego-Damia A, Macian-Gisbert V, Perpina-Tordera M, Roques-Serradilla JM. Maximal static respiratory pressures in children and adolescents. Pediatr Pulmonol. 2003 Feb;35(2):126-32. doi: 10.1002/ppul.10217. PMID 12526074
- [Background] Woszezenki CT, Heinzmann-Filho JP, Vendrusculo FM, Piva TC, Levices I, Donadio MV. Reference Values for Inspiratory Muscle Endurance in Healthy Children and Adolescents. PLoS One. 2017 Jan 25;12(1):e0170696. doi: 10.1371/journal.pone.0170696. eCollection 2017. PMID 28122012
- [Background] Beenakker EA, van der Hoeven JH, Fock JM, Maurits NM. Reference values of maximum isometric muscle force obtained in 270 children aged 4-16 years by hand-held dynamometry. Neuromuscul Disord. 2001 Jul;11(5):441-6. doi: 10.1016/s0960-8966(01)00193-6. PMID 11404114
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Uneri OS, Agaoglu B, Coskun A, Memik NC. Validity and reliability of Pediatric Quality of Life Inventory for 2- to 4-year-old and 5- to 7-year-old Turkish children. Qual Life Res. 2008 Mar;17(2):307-15. doi: 10.1007/s11136-007-9303-4. Epub 2008 Jan 18. PMID 18205028
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Background] Mahler DA, Rosiello RA, Harver A, Lentine T, McGovern JF, Daubenspeck JA. Comparison of clinical dyspnea ratings and psychophysical measurements of respiratory sensation in obstructive airway disease. Am Rev Respir Dis. 1987 Jun;135(6):1229-33. doi: 10.1164/arrd.1987.135.6.1229. PMID 3592398
- [Background] Ries AL, Bauldoff GS, Carlin BW, Casaburi R, Emery CF, Mahler DA, Make B, Rochester CL, Zuwallack R, Herrerias C. Pulmonary Rehabilitation: Joint ACCP/AACVPR Evidence-Based Clinical Practice Guidelines. Chest. 2007 May;131(5 Suppl):4S-42S. doi: 10.1378/chest.06-2418. PMID 17494825
- [Background] Tangye SG, Al-Herz W, Bousfiha A, Cunningham-Rundles C, Franco JL, Holland SM, Klein C, Morio T, Oksenhendler E, Picard C, Puel A, Puck J, Seppanen MRJ, Somech R, Su HC, Sullivan KE, Torgerson TR, Meyts I. Human Inborn Errors of Immunity: 2022 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2022 Oct;42(7):1473-1507. doi: 10.1007/s10875-022-01289-3. Epub 2022 Jun 24. PMID 35748970
- [Background] Kilic SS, Ozel M, Hafizoglu D, Karaca NE, Aksu G, Kutukculer N. The prevalences [correction] and patient characteristics of primary immunodeficiency diseases in Turkey--two centers study. J Clin Immunol. 2013 Jan;33(1):74-83. doi: 10.1007/s10875-012-9763-3. Epub 2012 Sep 15. PMID 22983506
- [Background] Ameratunga R, Longhurst H, Lehnert K, Steele R, Edwards ESJ, Woon ST. Are All Primary Immunodeficiency Disorders Inborn Errors of Immunity? Front Immunol. 2021 Jul 21;12:706796. doi: 10.3389/fimmu.2021.706796. eCollection 2021. No abstract available. PMID 34367167
- [Background] Hampson FA, Chandra A, Screaton NJ, Condliffe A, Kumararatne DS, Exley AR, Babar JL. Respiratory disease in common variable immunodeficiency and other primary immunodeficiency disorders. Clin Radiol. 2012 Jun;67(6):587-95. doi: 10.1016/j.crad.2011.10.028. Epub 2012 Jan 9. PMID 22226567
- [Background] Verma N, Grimbacher B, Hurst JR. Lung disease in primary antibody deficiency. Lancet Respir Med. 2015 Aug;3(8):651-60. doi: 10.1016/S2213-2600(15)00202-7. Epub 2015 Jul 15. PMID 26188881
- [Background] Modell V, Orange JS, Quinn J, Modell F. Global report on primary immunodeficiencies: 2018 update from the Jeffrey Modell Centers Network on disease classification, regional trends, treatment modalities, and physician reported outcomes. Immunol Res. 2018 Jun;66(3):367-380. doi: 10.1007/s12026-018-8996-5. PMID 29744770
- [Background] Quinti I, Di Pietro C, Martini H, Pesce AM, Lombardi F, Baumghartner M, Colantuono S, Milito C, Tabolli S. Health related quality of life in common variable immunodeficiency. Yonsei Med J. 2012 May;53(3):603-10. doi: 10.3349/ymj.2012.53.3.603. PMID 22477006
- [Background] Routes J, Costa-Carvalho BT, Grimbacher B, Paris K, Ochs HD, Filipovich A, Hintermeyer M, de Melo KM, Workman S, Ito D, Ye X, Bonnet P, Li-McLeod J. Health-Related Quality of Life and Health Resource Utilization in Patients with Primary Immunodeficiency Disease Prior to and Following 12 Months of Immunoglobulin G Treatment. J Clin Immunol. 2016 Jul;36(5):450-61. doi: 10.1007/s10875-016-0279-0. Epub 2016 Apr 18. PMID 27091140
- [Background] Urschel S, Kayikci L, Wintergerst U, Notheis G, Jansson A, Belohradsky BH. Common variable immunodeficiency disorders in children: delayed diagnosis despite typical clinical presentation. J Pediatr. 2009 Jun;154(6):888-94. doi: 10.1016/j.jpeds.2008.12.020. Epub 2009 Feb 23. PMID 19230900
- [Background] Jesenak M, Banovcin P, Jesenakova B, Babusikova E. Pulmonary manifestations of primary immunodeficiency disorders in children. Front Pediatr. 2014 Jul 25;2:77. doi: 10.3389/fped.2014.00077. eCollection 2014. PMID 25121077
- [Background] Azizi G, Abolhassani H, Asgardoon MH, Alinia T, Yazdani R, Mohammadi J, Rezaei N, Ochs HD, Aghamohammadi A. Autoimmunity in common variable immunodeficiency: epidemiology, pathophysiology and management. Expert Rev Clin Immunol. 2017 Feb;13(2):101-115. doi: 10.1080/1744666X.2016.1224664. Epub 2016 Sep 16. PMID 27636680
- [Background] Manson D, Reid B, Dalal I, Roifman CM. Clinical utility of high-resolution pulmonary computed tomography in children with antibody deficiency disorders. Pediatr Radiol. 1997 Oct;27(10):794-8. doi: 10.1007/s002470050235. PMID 9323243
- [Background] ERS Task Force; Palange P, Ward SA, Carlsen KH, Casaburi R, Gallagher CG, Gosselink R, O'Donnell DE, Puente-Maestu L, Schols AM, Singh S, Whipp BJ. Recommendations on the use of exercise testing in clinical practice. Eur Respir J. 2007 Jan;29(1):185-209. doi: 10.1183/09031936.00046906. PMID 17197484
- [Background] Clinical exercise testing with reference to lung diseases: indications, standardization and interpretation strategies. ERS Task Force on Standardization of Clinical Exercise Testing. European Respiratory Society. Eur Respir J. 1997 Nov;10(11):2662-89. doi: 10.1183/09031936.97.10112662. No abstract available. PMID 9426113
- [Background] Mattiello R, Sarria EE, Stein R, Fischer GB, Mocelin HT, Barreto SS, Lima JA, Brandenburg D. Functional capacity assessment in children and adolescents with post-infectious bronchiolitis obliterans. J Pediatr (Rio J). 2008 Jul-Aug;84(4):337-43. doi: 10.2223/JPED.1807. PMID 18688552
- [Background] Frohlich LF, Vieira PJ, Teixeira PJ, Silva FA, Ribeiro JP, Berton DC. Exercise capacity in adolescent and adult patients with post infectious bronchiolitis obliterans. Pediatr Pulmonol. 2014 Sep;49(9):911-8. doi: 10.1002/ppul.22929. Epub 2013 Dec 23. PMID 24375976
- [Background] Zenteno D, Puppo H, González R, Pavón D, Vera R, Torres R. Six minute walk test in children with post-infectious obliterans bronchiolitis. Its relation with spirometry. Rev Chil Enferm Respir. 2008;24:15-19. 24.
- [Background] Gerbase MW, Soccal PM, Spiliopoulos A, Nicod LP, Rochat T. Long-term health-related quality of life and walking capacity of lung recipients with and without bronchiolitis obliterans syndrome. J Heart Lung Transplant. 2008 Aug;27(8):898-904. doi: 10.1016/j.healun.2008.04.012. Epub 2008 Jun 10. PMID 18656804